CLINICAL TRIAL: NCT01165268
Title: Characterization of the Kinetics of Renal Glucose Reabsorption in Response to Dapagliflozin in Healthy Subjects and in Subjects With Type 2 Diabetes Mellitus
Brief Title: Characterization of the Kinetics of Renal Glucose Reabsorption in Response to Dapagliflozin in Healthy Subjects and in Subjects With Type 2 Diabetes Mellitus (T2DM)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: MB102-066
Record Dates: First submitted 2010-07-16; First posted 2010-07-19 (Estimated); Last update posted 2016-11-17 (Estimated); Status verified 2016-11

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dapagliflozin (T2DM) (Active Comparator)
  Interventions: Drug: Dapagliflozin
- Dapagliflozin (Healthy Subjects) (Active Comparator)
  Interventions: Drug: Dapagliflozin

INTERVENTIONS:
Drug: Dapagliflozin — Tablets, Oral, 10 mg, Once daily, 7 days

SUMMARY:
It is anticipated that 7 days of oral administration of 10 mg dapagliflozin will reduce the renal glucose reabsorption similarly in healthy subjects and in subjects with T2DM.

ELIGIBILITY:
Inclusion criteria for T2DM

* Diagnosis of T2DM
* Must be on one of the following therapies: diet therapy alone, diet plus a sulfonylurea, diet plus metformin, or diet plus sulfonylurea plus metformin
* Subjects taking metformin, and/or sulfonylurea must be on a stable dose for at least 2 months prior to study drug administration
* Must have a fasting plasma glucose concentration ≤ 200 mg/dl, and HbA1C ≤ 10%

Inclusion criteria for healthy subjects:

* Healthy subjects (as determined by no clinically significant deviation from normal in medical history, physical examination, ECGs, and clinical laboratory determinations)

Inclusion criteria for all subjects:

* Subjects with (eGFR ≥ 60 and ≤ 160 mL/min/1.73m² and urinary albumin excretion < 300 mg/g creatinine)
* Body Mass Index (BMI) of 18 to 38 kg/m²
* Men and women, ages 18 to 65 years, inclusive

Exclusion criteria for all subjects:

* Subjects with Type 1 Diabetes or uncontrolled Type 2 Diabetes Mellitus
* Subjects with T2DM with fasting plasma glucose > 200 mg/dL, healthy subjects with fasting plasma glucose > 105 mg/dL
* Subjects with T2DM with HbA1C > 10.0%, healthy subjects with HbA1C > 6.8%

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-08; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
The reduction in TmG after 7 days of oral administration of 10 mg of dapagliflozin | Before 7 days of oral administration of 10 mg of dapagliflozin
The reduction in TmG after 7 days of oral administration of 10 mg of dapagliflozin | After 7 days of oral administration of 10 mg of dapagliflozin

SECONDARY OUTCOMES:
Splay of the glucose titration curve | Before 7 days of oral administration of 10 mg of dapagliflozin
Splay of the glucose titration curve | After 7 days of oral administration of 10 mg of dapagliflozin
Pharmacokinetics (Cmin, Cmax, Tmax, and AUC (TAU)) of dapagliflozin | Study Day 7
Pharmacokinetics (Cmin, Cmax, Tmax, and AUC (TAU)) of dapagliflozin | Study Day 8

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Profil Institute For Clinical Research, Inc., Chula Vista, California, United States

REFERENCES:
- See also: MB102-066_CSR_synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3651&filename=MB102-066_CSR_synopsis.pdf